CLINICAL TRIAL: NCT00021502
Title: A Phase 3, Multi-Center, Randomized, Placebo Controlled Study of PHP When Administered by Continuous Infusion in Patients With Shock Associated With Systemic Inflammatory Response Syndrome (SIRS)
Brief Title: Safety and Efficacy of PHP in the Treatment of Shock Associated With Systemic Inflammatory Response Syndrome (SIRS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Apex Bioscience (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APX-PHP 99-004
Record Dates: First submitted 2001-07-18; First posted 2001-07-20 (Estimated); Last update posted 2009-08-14 (Estimated); Status verified 2009-08

CONDITIONS: Shock; Systemic Inflammatory Response Syndrome
Keywords: Pyridoxalated hemoglobin polyoxyethylene conjugate (PHP); Systemic Inflammatory Response Syndrome (SIRS); Nitric oxide (NO); Shock
MeSH Terms: conditions — Shock; Systemic Inflammatory Response Syndrome | interventions — pyridoxalated-hemoglobin-polyethylene glycol conjugate

INTERVENTIONS:
Drug: pyridoxalated hemoglobin polyoxyethylene conjugate (PHP)

SUMMARY:
To determine the safety and effectiveness of pyridoxylated hemoglobin polyoxyethylene conjugate (PHP) administered by continuous intravenous (IV) infusion in systemic inflammatory response syndrome (SIRS) patients with shock. PHP is a human-derived chemically modified hemoglobin preparation. PHP selectively scavenges excess nitric oxide (NO) and does so in a catalytic, concentration-dependent reaction that results in the formation of the non-toxic NO metabolite, nitrate. PHP is postulated to reduce excess, toxic levels of NO while allowing critical beneficial levels of the molecule to persist.

DETAILED DESCRIPTION:
This Phase 3, randomized, placebo controlled, multi-center study is designed to evaluate the safety and efficacy of continuous IV infusion of PHP plus conventional vasopressor treatment, as compared to continuous IV infusion of Plasma-Lyte A plus conventional vasopressor, as a treatment for restoring hemodynamic stability in SIRS patients with shock. Conventional vasopressors include dopamine > 5 mcg/kg/min; or norepinephrine, phenylephrine or epinephrine at any dose.

The study consists of a Screening period, a Pre-Treatment period, and a 28-day Treatment period. Efficacy will be determined by evaluating objective clinical measures of mortality and organ function over the 28-day treatment period.

The safety and tolerability of PHP will be evaluated over the continuous 28 days using a number of measures including an evaluation of:

* all cause mortality,
* median patient survival time and
* adverse event rates and duration.

ELIGIBILITY:
Determination of study eligibility will be made by the Investigator on the basis of the inclusion criteria listed below:

SIRS Inclusion Criteria

Patients with SIRS as characterized by two or more of the following conditions (worst values in a 24 hour period):

* Either respiratory rate >/= 20 breaths/minute, partial pressure of arterial carbon dioxide (PaCO2) </= 32 torr, or mechanical ventilation,
* Heart rate >/= 90 beats/minute,
* Either hyperthermia >/= 38 degrees C, or hypothermia </= 36 degrees C or
* Either white blood cell (WBC) >/= 12,000 cells/mm3, </= 4,000 cells/mm3, or >/= 10% immature (band) forms

Shock Inclusion Criteria Patients with adequate fluid resuscitation (PCWP >/= 12mmHg) and with one or more conventional vasopressors (continuing up to the time of randomization) being used to treat hypotension (MBP < 60 mmHg or SBP < 90 mmHg). Patients cannot be entered if they have been in shock for more than 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000
Dates: Start 2001-03; Primary Completion 2003-08 (Actual); Study Completion 2004-05 (Actual)

REFERENCES:
- [Result] Kinasewitz GT, Privalle CT, Imm A, Steingrub JS, Malcynski JT, Balk RA, DeAngelo J. Multicenter, randomized, placebo-controlled study of the nitric oxide scavenger pyridoxalated hemoglobin polyoxyethylene in distributive shock. Crit Care Med. 2008 Jul;36(7):1999-2007. doi: 10.1097/CCM.0b013e31817bfe84. PMID 18552688